CLINICAL TRIAL: NCT00281788
Title: A Phase I Study of Oral Capecitabine in Combination With Weekly IV Carboplatin/Paclitaxel and Radiation Therapy for Patients
Brief Title: Combination Chemotherapy and Radiation Therapy in Treating Patients With Esophageal Cancer or Gastroesophageal Junction Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: 4950; DUMC-4950-05-8R2; CDR0000449942 (Other: NCI)
Record Dates: First submitted 2006-01-24; First posted 2006-01-25 (Estimated); Last update posted 2013-03-21 (Estimated); Status verified 2008-04

CONDITIONS: Esophageal Cancer
Keywords: stage I esophageal cancer; stage II esophageal cancer; stage III esophageal cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Capecitabine; Carboplatin; Paclitaxel; Radiotherapy

INTERVENTIONS:
Drug: capecitabine
Drug: carboplatin
Drug: paclitaxel
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as capecitabine, carboplatin, and paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving chemotherapy together with radiation therapy may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of capecitabine when given together with carboplatin, paclitaxel, and radiation therapy in treating patients with esophageal cancer or gastroesophageal junction cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose and recommended phase II dose of capecitabine when administered with carboplatin, paclitaxel, and radiotherapy in patients with carcinoma of the esophagus or gastroesophageal junction.

Secondary

* Determine the radiographic and pathologic response rate in patients treated with this regimen.
* Correlate, preliminarily, tumor biomarker response with clinical response in patients treated with this regimen.

OUTLINE: This is an open-label, dose-escalation study of capecitabine.

Patients undergo radiotherapy once daily and receive oral capecitabine twice daily on days 1-5 and carboplatin IV over 30 minutes and paclitaxel IV over 1 hour on day 2. Treatment repeats weekly for 5 weeks in the absence of disease progression or unacceptable toxicity. Beginning at week 9 (4 weeks after completing chemoradiotherapy), some patients may undergo surgery to remove the tumor. Patients with unresectable or gross residual disease after completing radiotherapy may continue to receive capecitabine, carboplatin, and paclitaxel for as long as the chemotherapy is beneficial.

Cohorts of 3-6 patients receive escalating doses of capecitabine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity.

PROJECTED ACCRUAL: A total of 36 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed carcinoma of the thoracic esophagus or gastroesophageal junction for which bimodality treatment with chemotherapy and radiotherapy is indicated
* No tumors that extend above the level of the thoracic inlet or beyond 4 cm below the gastroesophageal junction
* No esophageal perforation based on radiographic or bronchoscopic evidence
* No known brain metastases, lymphangitic lung metastases, or carcinomatous meningitis

PATIENT CHARACTERISTICS:

* Karnofsky performance status ≥ 70%
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* AST or ALT ≤ 2.5 times upper limit of normal (ULN)
* Bilirubin ≤ 1.5 mg/dL
* Creatinine ≤ 1.5 times ULN
* Calcium ≤ 1.3 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No active infection or other serious underlying medical condition that would preclude study treatment
* No dementia or significantly altered mental status that would preclude understanding or giving informed consent

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy or radiotherapy
* No other concurrent investigational therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2003-09; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Herbert I. Hurwitz, MD, Principal Investigator — Duke Cancer Institute
Locations (1):
- Duke Comprehensive Cancer Center, Durham, North Carolina, United States